CLINICAL TRIAL: NCT01743521
Title: Direct Acting Antiviral (DAA) Based Therapy for Recently Acquired Hepatitis C
Brief Title: DAA Based Therapy for Recently Acquired Hepatitis C (DARE-C)
Acronym: DARE-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1102; VX-950HCP4010 (Other Grant/Funding Number: Janssen)
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Individualised therapy; Response-guided therapy; Telaprevir; PEG-IFN; Ribavirin; Hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A - 8 weeks total therapy (Experimental): 8 weeks total therapy of TPV/PEG-IFN/RBV if undetectable HCV RNA after 2 weeks of therapy
  Interventions: Drug: TPV/PEG-IFN/RBV
- Group B - 12 weeks total therapy (Experimental): 12 weeks total therapy of TPV/PEG-IFN/RBV if undetectable HCV RNA after 4 weeks of therapy
  Interventions: Drug: TPV/PEG-IFN/RBV
- Group C - 24 weeks total therapy (Experimental): 24 weeks total therapy - TPV/PEG-IFN/RBV for 12 weeks + PEG-IFN/RBV for 12 weeks if undetectable HCV RNA after 8 weeks of therapy
  Interventions: Drug: TPV/PEG-IFN/RBV

INTERVENTIONS:
Drug: TPV/PEG-IFN/RBV — Drug Telaprevir (TPV): dosed 1125mg twice daily (given as three 375 mg film-coated tablets) orally, except in the situation where a patient is on efavirenz in which case the dose of telaprevir will be 1125mg three times daily.
  Drug Ribavirin (RBV): 1000mg or 1200mg p.o daily in split doses (1000mg for patients weighing <75kg and 1200mg for patients weighing ≥ 75kg).
  Drug PEG-IFN (other name: Pegasys): 180mcg in 0.5ml (pre-filled syringes) administered subcutaneously once weekly.
  Other Names: Telaprevir brand name: INCIVO; Ribavirin brand name: COPEGUS; PEG-IFN brand name: PEGASYS

SUMMARY:
To examine the safety and efficacy of response guided triple therapy (PEG-IFN, Ribavirin, Telaprevir) for the treatment of early chronic Hepatitis C Virus (HCV) infection.

DETAILED DESCRIPTION:
DARE-C is a prospective open label multi-centre pilot study examining the safety and efficacy of response guided triple therapy (PEG-IFN, Ribavirin and Telaprevir) for the treatment of early chronic HCV genotype 1 infection in individuals with and without HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written, informed consent.
2. HCV genotype 1 infection
3. Quantifiable HCV RNA at screening and baseline (>10,000 IU/ml)
4. Recent hepatitis C infection with an estimated duration of Infection >6 months and ≤ 18 months defined as A) i) First anti-HCV antibody or HCV RNA positive within the previous 6 months and ii) Documented anti-HCV antibody negative or HCV RNA negative within the 24 months prior to anti-HCV antibody positive result OR B) i) First anti-HCV antibody or HCV RNA positive within the previous 6 months and ii) acute clinical hepatitis (jaundice or ALT> 10 X ULN) within the 12 months prior to first positive HCV antibody or HCV RNA with no other cause of acute hepatitis identifiable
5. Compensated liver disease (Child-Pugh A)
6. Negative pregnancy test at screening and 24 hours prior to the first dose of study drugs.
7. If heterosexually active, a female subject of childbearing potential and a nonvasectomized male subject who has a female partner of childbearing potential must agree to use 2 effective contraceptives from screening onwards until 6 months (female subject) or 7 months (male subject) after RBV therapy has ended. Note: Hormonal contraceptives may be continued but may not be reliable during telaprevir dosing and for 2 months following cessation of telaprevir. Therefore, subjects should agree to use 2 effective non-hormonal methods of contraception during telaprevir combination therapy and for 2 months after the last intake of telaprevir. As of two months after completion of telaprevir hormonal contraceptives can again be used as one of the two required effective methods of birth control.
8. Subject is judged to be medically stable on the basis of physical examination, medical history and vital signs.
9. Adequate English to provide written, informed consent and to provide reliable responses to the study interview

Additional inclusion criteria for HIV positive individuals

* Confirmed HIV infection > 6 months duration
* CD4 > 200 cells/mm3 and HIV < 50 c/ml on stable antiretroviral therapy (ART) at least 3 months prior to treatment
* Or
* CD4 >= 500 cells/mm3 and HIV viral load (VL) < 100,000 not on ART
* If on ART must be taking a regimen containing an accepted* combination of the following drugs: tenofovir ( TDF), lamivudine ( 3TC), emtricitabine (FTC), efavirenz (EFV), abacavir (ABC), raltegravir (RAL), etravirine (ETV), rilpivirine (RIL), ritonavir boosted atazanavir (r/ATZ) * Combination must be supported by current HIV treatment guidelines

Exclusion Criteria:

* Individuals considered by the study investigators to be unlikely to participate in intensive follow-up and/or unwilling to provide extra blood samples
* Current injecting drug use (any injecting within previous 4 weeks)
* Standard exclusions to Pegylated-interferon (PEG-IFN), Ribavirin (RBV) and Telaprevir (TPV) therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MbChB, PhD, Study Chair — Kirby Institute
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinello M, Hellard M, Shaw D, Petoumenos K, Applegate T, Grebely J, Yeung B, Maire L, Iser D, Lloyd A, Thompson A, Sasadeusz J, Haber P, Dore GJ, Matthews GV. Short duration response-guided treatment is effective for most individuals with recent hepatitis C infection: the ATAHC II and DARE-C I studies. Antivir Ther. 2016;21(5):425-34. doi: 10.3851/IMP3035. Epub 2016 Feb 11. PMID 26867206

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - 8 Weeks Total Therapy: 8 weeks total therapy of TPV/PEG-IFN/RBV if undetectable HCV RNA after 2 weeks of therapy
  TPV/PEG-IFN/RBV: Drug Telaprevir (TPV): dosed 1125mg twice daily (given as three 375 mg film-coated tablets) orally, except in the situation where a patient is on efavirenz in which case the dose of telaprevir will be 1125mg three times daily.
  Drug Ribavirin (RBV): 1000mg or 1200mg p.o daily in split doses (1000mg for patients weighing <75kg and 1200mg for patients weighing ≥ 75kg).
  Drug PEG-IFN (other name: Pegasys): 180mcg in 0.5ml (pre-filled syringes) administered subcutaneously once weekly.
- Group B - 12 Weeks Total Therapy: 12 weeks total therapy of TPV/PEG-IFN/RBV if undetectable HCV RNA after 4 weeks of therapy
  TPV/PEG-IFN/RBV: Drug Telaprevir (TPV): dosed 1125mg twice daily (given as three 375 mg film-coated tablets) orally, except in the situation where a patient is on efavirenz in which case the dose of telaprevir will be 1125mg three times daily.
  Drug Ribavirin (RBV): 1000mg or 1200mg p.o daily in split doses (1000mg for patients weighing <75kg and 1200mg for patients weighing ≥ 75kg).
  Drug PEG-IFN (other name: Pegasys): 180mcg in 0.5ml (pre-filled syringes) administered subcutaneously once weekly.
- Group C - 24 Weeks Total Therapy: 24 weeks total therapy - TPV/PEG-IFN/RBV for 12 weeks + PEG-IFN/RBV for 12 weeks if undetectable HCV RNA after 8 weeks of therapy
  TPV/PEG-IFN/RBV: Drug Telaprevir (TPV): dosed 1125mg twice daily (given as three 375 mg film-coated tablets) orally, except in the situation where a patient is on efavirenz in which case the dose of telaprevir will be 1125mg three times daily.
  Drug Ribavirin (RBV): 1000mg or 1200mg p.o daily in split doses (1000mg for patients weighing <75kg and 1200mg for patients weighing ≥ 75kg).
  Drug PEG-IFN (other name: Pegasys): 180mcg in 0.5ml (pre-filled syringes) administered subcutaneously once weekly.
- No Group Allocated: Early treatment discontinuation or non-responder (participants in whom therapy was terminated at week 4 due to HCV RNA >1000 IU/mL or week 8 due to detectable HCV RNA)
Period: Overall Study
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy | No Group Allocated
Started | 7 | 3 | 2 | 2
Completed | 7 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Group Allocated: Early treatment discontinuation or non-responder
- Total: Total of all reporting groups
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy | No Group Allocated | Total
Number analyzed (Participants) | 7 | 3 | 2 | 2 | 14
Age, Continuous [Median (Full Range); unit: years] | 49 [28 to 65] | 45 [35 to 49] | 44 [33 to 54] | 57 [46 to 68] | 48 [28 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 3 | 2 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 3 | 2 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Estimated Duration of infection at baseline [Median (Inter-Quartile Range); unit: weeks] | 39 [25 to 56] | 46 [36 to 75] | 50 [41 to 59] | 33 [24 to 41] | 40.9 [36.4 to 56.4]
HIV infection [Number; unit: participants] | 5 | 2 | 2 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: SVR12 (Sustain Virological Response, HCV RNA Undetectable 12 Weeks Post-treatment)
Description: Proportion of subjects achieving SVR 12 (negative qualitative HCV RNA 12 weeks after therapy completion)
Time Frame: 12 weeks post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
percentage of participants | 71 | 100 | 100

2. Secondary Outcome: SVR24
Description: To evaluate the proportion of patients with undetectable HCV RNA 24 weeks after therapy completion (SVR24)
Time Frame: 24 weeks post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
percentage of participants | 43 | 100 | 100

3. Secondary Outcome: Undetectable HCV RNA (ETR)
Description: To evaluate the proportion of patients with undetectable HCV RNA at end of treatment (ETR)
Time Frame: Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
percentage of participants | 100 | 100 | 100

4. Secondary Outcome: Undetectable HCV RNA (Week 1)
Description: To evaluate the proportion of patients with undetectable HCV RNA at week 1 of therapy.
Time Frame: Week 1 of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
percentage of participants | 71.43 | 0 | 0

5. Secondary Outcome: Undectectable HCV RNA (Week 2)
Description: To evaluate the proportion of patients with undetectable HCV RNA at week 1 of therapy.
Time Frame: Week 2 of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
percentage of participants | 100 | 0 | 0

6. Secondary Outcome: Undetectable HCV RNA (Week 3)
Description: To evaluate the proportion of patients with undetectable HCV RNA at week 3 of therapy.
Time Frame: Week 3 of therapy
Population: Missing data carried forward if previously <LLoQ (lower limit of quantification)
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 5 | 2 | 2
percentage of participants | 100 | 33.33 | 0

7. Secondary Outcome: Undetectable HCV RNA (Week 4)
Description: To evaluate the proportion of patients with undetectable HCV RNA at week 4 of therapy.
Time Frame: Week 4 of therapy
Population: Missing data carried forward if previously <LLoQ
Measure: Number; unit: percentage of participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 5 | 3 | 2
percentage of participants | 100 | 66.67 | 0

8. Secondary Outcome: Decrease in Absolute Neutrophil Count (ANC) ≤0.75
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Measure: Number; unit: participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
participants | 1 | 1 | 0

9. Secondary Outcome: Decrease in Platelets <50
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Measure: Number; unit: participants
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
participants | 0 | 0 | 0

10. Secondary Outcome: Change in Hemoglobin at End of Treatment
Description: To evaluate indicators of toxicity during telaprevir based therapy
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 7 | 3 | 2
g/L | -31 [-43 to -15] | -53 [-63 to -47] | -17.5 [-21 to -14]

11. Secondary Outcome: Resistance-associated Variants
Description: To examine the emergence of resistance-associated variants during telaprevir based therapy for early chronic infection
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Population: Resistance-associated variants analysis have not yet been performed. These are planned to be performed at a later date.
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Baseline Resistance-associated Variants
Description: To correlate the presence and frequency of baseline resistance-associated variants (RAVs) with the response of Telaprevir based therapy for early chronic HCV infection.
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Population: Baseline resistance-associated variants analysis have not yet been performed. These are planned to be performed at a later date.
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Plasma Ribavirin Levels
Description: To correlate plasma ribavirin levels with treatment outcome and changes in haemoglobin during therapy
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Population: Ribavirin concentration have not yet been performed. These are planned to be performed at a later date.
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: CD4 and HIV RNA
Description: In HIV positive participants to evaluate changes in CD4 counts and HIV RNA during telaprevir based therapy
Time Frame: Baseline, Wk 8 (Group A), Wk 12 (Group B), Wk 24 (Group C)
Population: This data will not be analysed.
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Gene IL28B Polymorphism
Description: To examine treatment outcome by IL28B polymorphism
Time Frame: Baseline
Population: IL28B polymorphisms have not yet been performed. These are planned to be performed at a later date.
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events encountered during treatment and for 24 weeks after treatment discontinuation were reported for each participant.
Arm/Group | Group A - 8 Weeks Total Therapy | Group B - 12 Weeks Total Therapy | Group C - 24 Weeks Total Therapy
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - 8 Weeks Total Therapy (N=7) | Group B - 12 Weeks Total Therapy (N=3) | Group C - 24 Weeks Total Therapy (N=2)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Axillary Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - 8 Weeks Total Therapy (N=7) | Group B - 12 Weeks Total Therapy (N=3) | Group C - 24 Weeks Total Therapy (N=2)
Fatigue (General disorders) | 4 (4) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2) | 2 (2)
Change in mood (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Perianal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Irritability (General disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No